CLINICAL TRIAL: NCT00745316
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Assess the Safety and Tolerability of Oral Tonapofylline in Patients With Heart Failure and Renal Insufficiency
Brief Title: Oral Tonapofylline (BG9928) in Patients With Heart Failure and Renal Insufficiency
Acronym: POSEIDON
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company Decision
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 161HF201
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Renal Insufficiency; Heart Failure
Keywords: Heart Failure; Renal Insufficiency; Congestive Heart Failure
MeSH Terms: conditions — Renal Insufficiency; Heart Failure | interventions — BG 9928

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental): oral Dose 1
  Interventions: Drug: Tonapofylline
- 2 (Experimental): oral Dose 2
  Interventions: Drug: Tonapofylline
- 3 (Experimental): oral Dose 3
  Interventions: Drug: Tonapofylline
- 4 (Experimental): oral Dose 4
  Interventions: Drug: Tonapofylline
- 5 (Experimental): oral Dose 5
  Interventions: Drug: Tonapofylline
- 6 (Placebo Comparator): Placebo - 2 capsules bid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tonapofylline — Oral Tonapofylline - 2 capsules bid
  Other Names: BG9928; Selective Adenosine A1 Receptor Antagonist
  Arms: 1; 2; 3; 4; 5
Drug: Placebo — Oral placebo - 2 capsules bid
  Arms: 6

SUMMARY:
The main purpose of this study is to determine the safety and tolerability of tonapofylline (BG9928) when given at different doses to patients with heart failure and renal insufficiency.

This study will also explore:

* Disease related quality-of-life
* Exercise capacity
* Renal function
* Concomitant medications

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Diagnosis of heart failure requiring hospitalization >1 and ≤12 months prior to screening
* NYHA Class III or IV at the time of screening
* Renal insufficiency as defined by eGFR ≥20 and ≤70 mL/min/1.73 m2
* Negative pregnancy test

Exclusion Criteria:

* History of an allergic reaction to any xanthine-containing compound.
* History of seizure
* History of stroke
* Serious systemic infection
* Sustained systolic blood pressure >170 or <90 mmHg
* Myocardial infarction within 30 days of Day 1
* Hemodynamically destabilizing arrhythmia within 30 days of Day 1
* Uncorrected hemodynamically significant primary valvular disease
* Known obstructive or restrictive cardiomyopathy
* Cardiac surgery within 60 days prior to Day 1
* Likely to undergo cardiac transplantation, device implantation, or other cardiac surgery within next three months
* Evidence of malignancy within 6 months prior to Day 1.
* Participation in any other investigational study of drugs or devices within 30 days prior to Day 1.
* Receiving aminophylline, theophylline, pentoxifylline, dyphylline or adenosine
* Presence of any clinically significant condition that might interfere with optimal safe participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability of BG9928 administered to subjects with heart failure and renal insufficiency. | 16 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (28):
- United States (28):
  - Huntsville, Alabama
  - Mobile, Alabama
  - Scottsdale, Arizona
  - Tucson, Arizona
  - Beverly Hills, California
  - San Diego, California
  - Denver, Colorado
  - Bridgeport, Connecticut
  - Jacksonville, Florida
  - Melbourne, Florida
  - Ormond Beach, Florida
  - Chicago, Illinois
  - Maywood, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Owensboro, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Minneapolis, Minnesota
  - Lincoln, Nebraska
  - The Bronx, New York
  - Cincinnati, Ohio
  - Oklahoma City, Oklahoma
  - Lancaster, Pennsylvania
  - Germantown, Tennessee
  - Roanoke, Virginia
  - Beloit, Wisconsin
  - Madison, Wisconsin